CLINICAL TRIAL: NCT01174732
Title: Phase II Study Randomized, Double- or Evaluator-blind, Active- and Placebo-controlled, Single Dose, Seven-arm, Cross-over and Dose-ranging Study of A006 DPI, Albuterol Inhalation Powder, in Adult Asthma Patients
Brief Title: Dose-Ranging Study of A006 DPI, in Adult Asthma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: API-A006-CL-B
Record Dates: First submitted 2010-07-29; First posted 2010-08-04 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Asthma; Bronchospasm
Keywords: asthma; bronchospasm; COPD; chronic respiratory disease
MeSH Terms: conditions — Asthma; Bronchial Spasm; Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- T1 (Experimental): A006 albuterol inhalation powder, 120 mcg/inhalation, 1 inhalation
  Interventions: Drug: albuterol inhalation powder
- T2 (Experimental): A006 albuterol inhalation powder 180 mcg/ inhalation, 1 inhalation
  Interventions: Drug: albuterol inhalation powder
- T3 (Experimental): A006 albuterol inhalation powder, 120 mcg/inhalation, 2 inhalations
  Interventions: Drug: albuterol inhalation powder
- T4 (Experimental): A006 albuterol inhalation powder 180 mcg/inhalation, 2 inhalations
  Interventions: Drug: albuterol inhalation powder
- P (Placebo Comparator): Placebo, 2 inhalations
  Interventions: Drug: Placebo
- R1 (Active Comparator): Proventil 90 mcg/inhalation, 2 inhalations
  Interventions: Drug: albuterol inhalation aerosol
- R2 (Active Comparator): Proventil 90 mcg/inhalation, 4 inhalations
  Interventions: Drug: albuterol inhalation aerosol

INTERVENTIONS:
Drug: albuterol inhalation powder — A006 albuterol inhalation powder, 120 mcg/inhalation, one inhalation
  Arms: T1
Drug: albuterol inhalation powder — A006 albuterol inhalation powder, 180 mcg/inhalation, 1 inhalation
  Arms: T2
Drug: albuterol inhalation powder — A006 albuterol inhalation powder, 120 mcg/inhalation, 2 inhalations
  Arms: T3
Drug: albuterol inhalation powder — A006 albuterol inhalation powder, 180 mcg/inhalation, 2 inhalations
  Arms: T4
Drug: Placebo — placebo, lactose inhalation carrier
  Arms: P
Drug: albuterol inhalation aerosol — albuterol inhalation aerosol, 90 mcg/inhalation, 2 inhalations
  Other Names: Proventil
  Arms: R1
Drug: albuterol inhalation aerosol — albuterol inhalation aerosol, 90 mcg/inhalation, 4 inhalations
  Other Names: Proventil
  Arms: R2

SUMMARY:
This study is a randomized, active- and placebo-controlled, single-dose, seven-arm, crossover and dose-ranging design. This study aims to evaluate the efficacy and initial safety profiles, and to identify the optimum dose of A006, from a select dose-range for future clinical PK/PD and Phase III studies. This study is to be conducted in generally healthy, adult subjects who have mild-to-moderate persistent asthma for at least 6 months prior to Screening.

ELIGIBILITY:
Inclusion Criteria:

* With mild-to-moderate persistent asthma for at least 6 months and having used inhaled beta-agonist for asthma control;
* Must demonstrate response to beta 2 agonist by Reversing;
* Must demonstrate ability to use DPI;
* Females of child-bearing potential must be non-pregnant, non-lactating, and practicing a clinically acceptable form of birth control;
* Additional Criteria

Exclusion Criteria:

* Smoking history of ≥ 10 pack-years, or having smoked within 6 months;
* Upper respiratory tract infections
* Asthma exacerbations;
* Known intolerance or hypersensitivity to any of the ingredients of the study drug or Proventil®;
* Use of prohibited drugs or failure to observe the drug washout restrictions;
* Having been on other clinical drug/device studies in the last 30 days;
* Other Criteria

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
AUC | 5, 20, 40, 60, 90; 120, 180, 240, and 360 minutes post-dose.
  Area under the curve (AUC) of post-dose FEV1 percentage changes from the Pre-dose Baseline. The primary analysis of the primary endpoint is to compare the AUC0-t of FEV1, between the A006 treatments and the Placebo Control.

SECONDARY OUTCOMES:
Time to Effect | 0 to 360 minutes
  Time to onset of bronchodilator effect
Peak Response | 0 - 360 minutes
  peak bronchodilator response
Duration | 0 - 360 minutes
  Duration of effect
Response Rate | 0 - 360 minutes
  Bronchodilatory Response Rate
Hand Tremor | within 5 min. prior to dosing and 50 and 360 min post-dose.
  Evaluation of hand tremor
Vital Signs | within 15 min. prior to dosing, and 30, 90 and 360 min post-dose.
  Pulse, heartrate, respirations, blood pressure
12 lead ECG | within 15 min. prior to dosing and at 50 and 360 min postdose.
  12-lead ECG for routine and QT/QTc evaluations
Blood Work | within 15 min. prior to dosing, and 30 and 120 min. postdose
  Collect blood samples (~5 mL) for serum glucose and K+ tests

CONTACTS AND LOCATIONS:
Overall Officials: Safety Monitor, Study Director — Amphastar Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Amphastar Site 0001, San Jose, California
  - Amphastar Site 0007, Centennial, Colorado
  - Amphastar Site 0008, Denver, Colorado
  - Amphastar Site 0039, Lakewood, Colorado